CLINICAL TRIAL: NCT05667259
Title: Prognostic Significance of Lymph Node Ratio in Rectal Cancer on Overall Survival: An Alternative Not a Substitute
Brief Title: Prognostic Significance of Lymph Node Ratio in Rectal Cancer on Overall Survival
Status: Completed | Type: Observational
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Abdallah Mohamed Taha Aly, Associate professor of General Surgry, South Valley University
Other Study IDs: SVU-MED-SUR011-4-22-10-464
Record Dates: First submitted 2022-12-19; First posted 2022-12-28 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Cancer, Rectum
Keywords: Cancer Rectum; Lymph node ratio; Overall Survival; Prognosis
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Surgical resection for cancer rectum — Curative resection for cancer recum

SUMMARY:
This study was conducted to compare the significance of lymph node ratio and absolute count of positive lymph node count on overall survival in patients with rectal cancer who underwent resection with curative intent

DETAILED DESCRIPTION:
Retrospective cohort study carried on 229 patients with non-metastatic rectal cancer, admitted in tertiary hospitals along 10 years, between 2012 to 2022, and underwent radical resection surgery with curative intent.

Exclusion criteria included patients with familial adenomatous polyposis, multiple synchronous or metachronous rectal cancers, early post-operative recurrence or death within 3 months. Demographic, histopathological, follow up and outcome data were collected.

Demographics included age, gender, family history, and chief complaint at presentation. Histopathological data included tumor site, grade, vascular-perineural invasion, total number of lymph nodes removed, and positive lymph nodes.

Lymph node ratio was defined as the ratio of positive lymph nodes to the total number of retrieved lymph nodes in histopathology specimen. Survival was calculated for each patient based on time of surgery to time of death

Statistical analysis will be used to evaluate the effect of lymph node ratio on overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Patient with rectal cancer of stage I-III.
* patients underwent radical resection with curative intent.

Exclusion Criteria:

* Patients with Familial Adenomatous Polyposis, multiple synchronous or metachronous rectal cancers.
* Early post-operative recurrence, or death within 3 months.

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with rectal cancer that were admitted in tertiary hospitals and underwent curative rectal resection. Patients' files were reviewed, and the data were collected and tabulated.
Sampling Method: Probability Sample
Enrollment: 229 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Overall Survival | up to 10 years (From date of surgery to the date date of death)
  Survival was calculated for each patient based on time of surgery to time of death.

CONTACTS AND LOCATIONS:
Overall Officials: Abdallah M Taha, MD, Principal Investigator — Egypt, South Valley University, Faculty of Medicine
Locations (1):
- Qena Faculty of Medicine, South Valley University Hospitals, Qina, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li Destri G, Di Carlo I, Scilletta R, Scilletta B, Puleo S. Colorectal cancer and lymph nodes: the obsession with the number 12. World J Gastroenterol. 2014 Feb 28;20(8):1951-60. doi: 10.3748/wjg.v20.i8.1951. PMID 24587671
- [Background] Amin MB, Greene FL, Edge SB, Compton CC, Gershenwald JE, Brookland RK, Meyer L, Gress DM, Byrd DR, Winchester DP. The Eighth Edition AJCC Cancer Staging Manual: Continuing to build a bridge from a population-based to a more "personalized" approach to cancer staging. CA Cancer J Clin. 2017 Mar;67(2):93-99. doi: 10.3322/caac.21388. Epub 2017 Jan 17. PMID 28094848
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Le Voyer TE, Sigurdson ER, Hanlon AL, Mayer RJ, Macdonald JS, Catalano PJ, Haller DG. Colon cancer survival is associated with increasing number of lymph nodes analyzed: a secondary survey of intergroup trial INT-0089. J Clin Oncol. 2003 Aug 1;21(15):2912-9. doi: 10.1200/JCO.2003.05.062. PMID 12885809
- [Background] Tepper JE, O'Connell MJ, Niedzwiecki D, Hollis D, Compton C, Benson AB 3rd, Cummings B, Gunderson L, Macdonald JS, Mayer RJ. Impact of number of nodes retrieved on outcome in patients with rectal cancer. J Clin Oncol. 2001 Jan 1;19(1):157-63. doi: 10.1200/JCO.2001.19.1.157. PMID 11134208